CLINICAL TRIAL: NCT04453371
Title: Tissue Plasminogen Activator (tPA) Treatment for an Atypical Acute Respiratory Distress Syndrome (Microvascular COVID-19 Lung Vessels Obstructive Thromboinflammatory Syndrome (MicroCLOTS): A Multicentral Randomized Trial (AtTAC-trial)
Brief Title: Impact of Tissue Plasminogen Activator (tPA) Treatment for an Atypical Acute Respiratory Distress Syndrome (COVID-19)
Acronym: AtTAC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Our local committee has denied the approval request
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Collaborators: Demikhov Municipal Clinical Hospital 68 (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tPA-2020
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: COVID-19; MicroCLOTS; Atypical Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Tissue Plasminogen Activator; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Thrombolysis
  Interventions: Drug: Tissue plasminogen activator
- Control group (Placebo Comparator): Ringer's solution infusion
  Interventions: Drug: Ringer solution

INTERVENTIONS:
Drug: Tissue plasminogen activator — In the study group, tPA (Alteplase) 25 mg i/v over 2 hours, followed by a 25 mg tPA infusion over the subsequent 22 hours. After the end of thrombolytic therapy, unfractionated heparin is administered i/v at a starting dose of 10 units / kg per hour. The target value of PTT is 40C-50C.
  In both groups patient's transfer from the heparin infusion to the introduction of low-molecular-weight heparins is performed after normalization of the D-dimer level.
  Other Names: Alteplase
  Arms: Study group
Drug: Ringer solution — In the control group, an equivalent amount of Ringer's solution is administered. After 24 hours, the heparin infusion gets started, similar the described for study group.
  In both groups patient's transfer from the heparin infusion to the introduction of low-molecular-weight heparins is performed after normalization of the D-dimer level.
  Arms: Control group

SUMMARY:
At the beginning COVID-associated lung injury was considered as typical ARDS, hence respiratory and nonrespiratory treatments were delivered according to general principles for this kind of illness. There is hypothesis that in predisposed individuals, alveolar viral damage is followed by an inflammatory reaction and by microvascular pulmonary thrombosis. The investigators suggest that thrombolytic therapy may be beneficial when compared to standard care in patients with SARS-CoV-2 and severe respiratory failure.

DETAILED DESCRIPTION:
COVID 19 pandemic is a serious challenge for International medical community. There is lack of knowledge about the nature and character of the lung injury caused by this kind of infection. At the beginning COVID-associated lung injury was considered as typical ARDS, hence respiratory and nonrespiratory treatments were delivered according to general principles for this kind of illness. There is hypothesis that in predisposed individuals, alveolar viral damage is followed by an inflammatory reaction and by microvascular pulmonary thrombosis. This progressive endothelial thromboinflammatory syndrome may also involve the microvascular bed of the brain and other vital organs, leading to multiple organ failure and death. Understanding the crucial role of microthrombosis in the genesis of SARS-2-CoV led to a widespread anticoagulant use. Moreover, there is evidence about a possible benefit of thrombolysis in patients with severe COVID-19 pulmonary disease. For Instance, some investigators reported about three patients with COVID 19 lung injury treated with alteplase (tPA). Authors oversaw positive changes in P/F ratio in 3/3 patients, even if in two of these patients changes lasted for a short period. Another investigators reported about the improvements in alveolar ventilation, arterial oxygenation and diminishing in vasopressor's support in 4 patients with SARS-2CoV after thrombolysis. Encouraging results were obtained also by another team in case series of 5 patients who received alteplase. Thus, there is evidence suggesting that thrombolytic therapy may be beneficial when compared to standard care in patients with SARS-CoV-2 and severe respiratory failure. This hypothesis is based on a well-established pathophysiological concept of the occurrence of pulmonary damage as a result of microthrombosis of the lung vessels. Hence, it seems crucial to conduct a randomized clinical trial to test the effectiveness of this treatment.

Objective: To establish whether plasminogen activator (tPA) treatment improves alveolar ventilation P/F (PaO2/FiO2) ratio will be calculated each 6 hours during first 3 days after the end of thrombolysis procedure in patients with an Atypical Acute Respiratory Distress Syndrome (Microvascular COVID-19 Lung Vessels Obstructive Thromboinflammatory Syndrome (MicroCLOTS).

Methods: Research assistants and/or clinician screen all mechanically ventilated patients for eligibility. Patients satisfying all of the Inclusion and Exclusion Criteria are classified as 'Eligible'. With informed consent from a substitute decision maker or under the decision of Concilium of three independent physicians, Eligible patients are 'Enrolled' into the study. Eligible patients Qualify for Randomization to one of the 2 groups: with or without thrombolytic therapy. In summary, patients are consented and Enrolled prior to Randomization. To enroll or randomize Eligible patients, research coordinators obtain informed consent and access the automated web-based system through Internet based program (available 24 hours/day). Each participating center has a separate computer-generated randomization schedule, with 1:1 (control to intervention) assignment, stratified by center, and using random variable block sizes.

The thrombolysis procedure: In the study group, tPA (Alteplase) 25 mg i/v over 2 hours, followed by a 25 mg tPA infusion over the subsequent 22 hours. After the end of thrombolytic therapy, unfractionated heparin is administered i/v at a starting dose of 10 units / kg per hour. The target value of PTT is 40C-50C. In the control group, an equivalent amount of Ringer's solution is administered. After 24 hours, the heparin infusion gets started, similar the described for study group.

In both groups patient's transfer from the heparin infusion to the introduction of low-molecular-weight heparins is performed after normalization of the D-dimer level.

Statistical analysis: Primary data analysis will be based on intention to treat (ITT) analysis.

Data will be analyzed also on a modified ITT approach (mITT). Will be included in this analysis only patients with evidence of an Atypical Acute Respiratory Distress Syndrome (Microvascular COVID-19 Lung Vessels Obstructive Thromboinflammatory Syndrome (MicroCLOTS).

Subgroups analysis: Some pre-defined subgroups analysis will be performed:

1. Patients with with P/F <200 mmHg>100 mmHg;
2. Patients with with P/F <100 mmHg;
3. Patient 65+ group;
4. Patients under 65 years old. Interim analyses: Interim analyses will not be performed

ELIGIBILITY:
Inclusion Criteria:

1. Severe pulmonary coronavirus disease 19 (COVID 19) with suspect for MicroCLOTS (microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome)
2. P/F ratio <200 mmHg> 70 mmHg
3. a.) Contrast CT scan positive for pulmonary thrombosis, OR b.) Contrast CT scan negative for pulmonary thrombosis:

   * D-Dimer > 10 mcg/mL, OR
   * 5 < D-dimer < 10 mcg/mL and C Reactive Protein (CRP) > 100 mg/dL

Exclusion Criteria:

* Age < 18
* Pregnancy or breastfeeding
* Known allergy to iodinated contrast dye
* Severe vasoplegic shock: norepinephrine > 300 ng/kg*min
* Glomerular Filtration rate < 30 ml/min
* Active bleeding or absolute contraindication to anticoagulant therapy (Stroke (intracranial hemorrhage, hemorrhagic stroke), including a history of the last 6 months.; cancer of the Central nervous system and other localities with an increased risk of bleeding, vascular aneurysm, traumatic open heart massage, obstetric delivery, General operations, severe uncontrolled hypertension, gastric ulcer and 12-duodenal ulcer (for 3 months. from the moment of exacerbation), arterial or venous malformations, liver failure, liver cirrhosis, portal hypertension, esophageal varicose veins, active hepatitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
P/F (PaO2/FiO2) change during the first 72hrs after the end of the procedure in adult patients with severe atypical ARDS caused by SARS-2-CoV. | Each 6 hours during first 3 days after the end of thrombolysis procedure.

SECONDARY OUTCOMES:
Ventilator-free time (days free from MV) for 28 days of observation. | 28 days
  Calculated as 28 days - number of days when patient receive any kind of ventilatory support (MV + SV + NIV).

OTHER OUTCOMES:
Mortality in 28 days and 1 year after randomization despite of the reason. | 28 days, 1 year after randomization
Length of stay in the ICU | 28 days
  Number of days when patient was in ICU
Length of stay in hospital | 28 days
  Number of days when patient was in hospital
The time needed for "improvement of 2 points" according to WHO "Ordinal Scale for Clinical Improvement" | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month
Chest radiographs on a daily basis and define barotrauma as the presence of new pneumothorax, pneumomediastinum, pneumoperitoneum, or subcutaneous emphysema. | Daily up to extubation than once a week/or on attending intensivist's discretion up to 1 month
Blood Pressure in millimetres of mercury | Each 4 hours during first 2 weeks after the end of thrombolysis procedure.
Heart Rate in beats per minute | Each 4 hours during first 2 weeks after the end of thrombolysis procedure.
Blood Oxygen Saturation | Each 4 hours during first 2 weeks after the end of thrombolysis procedure.
ECG Q-wave | Each 24 hours during first 2 weeks after the end of thrombolysis procedure.
ECG ST-segment | Each 24 hours during first 2 weeks after the end of thrombolysis procedure.